CLINICAL TRIAL: NCT03125330
Title: The Impact of Professional Coaching on Early Career Academic Emergency Physician Well-Being, Burnout, Leadership Strengths, and Goal Attainment: A Pilot Randomized, Controlled Trial
Brief Title: The Impact of Professional Coaching on Early Career Academic Emergency Physicians
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Richard C Winters, MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 16-010192
Record Dates: First submitted 2017-04-12; First posted 2017-04-24 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Development, Human; Well-Being; Professional Burnout; Goals; Leadership; Professional Role; Physician's Role; Stress; Anxiety
Keywords: Coaching; Professional coaching; Emergency physicians; Emergency medicine; Goal attainment; Leadership strengths; Well-being; Burnout; Adult level of development; Group coaching; Instructor; Assistant professor; Academic faculty; Subject-Object Interview
MeSH Terms: conditions — Burnout, Professional; Anxiety Disorders; Burnout, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- One-to-One Coaching (Experimental): Participants randomized to One-to-One Coaching meet for an initial 2-hour coaching session, followed by seven 1-hour coaching sessions every 3-weeks. These eight sessions take place over the course of 6 months.
  Additional requirements for One-to-One Coaching:
  * Complete a 30-minute online assessment of goal attainment, well-being, burnout, and leadership strengths (a) at study enrollment, (b) at 6-months after study enrollment, and (c) 12-months following study enrollment.
  * Complete a 15-minute VIA Character Strengths Test online prior to One-to-One Coaching.
  * Following the completion of the final coaching session, participants are interviewed by a con-investigator by phone call to assess the experience of coaching.
  Each coaching session will be recorded, transcribed, anonymized, and analyzed to identify common themes.
  Interventions: Behavioral: Professional coaching
- Group Coaching (Active Comparator): Participants meet for 90-minutes each month for 6 months for facilitated professional coaching with a group of colleagues.
  Additional requirements:
  * Complete a 30-minute online assessment of goal attainment, well-being, burnout, and leadership strengths (a) at study enrollment, (b) at 6-months after study enrollment, and (c) 12-months following study enrollment.
  * Complete a 15-minute VIA Character Strengths Test online prior to Group Coaching.
  * Prior to your initial group coaching session, participate in a 75-minute private phone interview with the primary investigator to discuss the how you make decisions and make sense of the world.
  * Following the completion of the final coaching session, participants are interviewed by a con-investigator by phone call to assess the experience of coaching.
  Each coaching session will be recorded, transcribed, anonymized, and analyzed to identify common themes.
  Interventions: Behavioral: Professional coaching
- Group Coaching Waitlist (No Intervention): Participants are offered group coaching at the completion of the 12-month study period. Six 90-minute group coaching sessions will occur over the course of six months.
  Additional requirements:
  • Complete a 30-minute online assessment of goal attainment, well-being, burnout, and leadership strengths (a) at study enrollment (b) and at 6-months after study enrollment.

INTERVENTIONS:
Behavioral: Professional coaching — Professional coaching is provided by the Principal Investigator via video conference.
  Other Names: Coaching
  Arms: Group Coaching; One-to-One Coaching

SUMMARY:
This research study is designed to answer the question: How does professional coaching impact early career academic emergency medicine physician goal attainment, leadership strengths, well-being, and burnout?

DETAILED DESCRIPTION:
A recent systematic review and meta-analysis found coaching to have significant positive effects on goal attainment, well-being, coping skills, work attitudes, and goal-directed self-regulation. Randomized controlled studies of professional coaching have found significant positive effects in various settings including high school teachers and students, postgraduate students in a major university, and executives in the commercial, government, and education sectors.

Coaching provides the participant focused time with a trained professional who facilitates that participant's self-determined and self-directed problem-solving and change. Coaching helps the participant "get on the balcony" away from the action on the "dance floor" to see things from a different and broader perspective and, in doing so, enriches the participant's ability to generate options, challenge biases, understand the effects of emotions, and consider uncertainty.

This study also establishes the level of adult development of academic faculty and creates an initial qualitative dataset for further longitudinal study and theory generation for physician well-being, burnout, leadership strengths, and goal attainment.

ELIGIBILITY:
Inclusion:

* Emergency physicians
* Academic appointment of Instructor or Assistant Professor
* Work greater than 80% of their time in a residency and fellowship program approved by the Accreditation Council of Graduate Medical Education (ACGME), the American Osteopathic Association (AOA), or the Royal College of Physicians and Surgeons of Canada (RCPSC) will be invited to participate in the study.

Exclusion:

* Mayo Clinic emergency physicians are not eligible for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2020-03-05 (Actual)

PRIMARY OUTCOMES:
Goal Setting and Attainment | 18 months (3 measurements at 6-month intervals)
  Each participant identifies two professional goals at study onset. For each of the goals, participants respond to the question, "Up to today, how successful have you been in achieving this goal?" and rate their goal attainment on a scale from 0% (no attainment) to 100% (complete attainment). To control for differences between participants in perceived goal attainment difficulty, participants also will rate each goal for perceived difficulty on a 4-point scale ( 1=very easy, 2=somewhat easy, 3=somewhat difficult, 4=very difficult). Goal attainment scores are calculated by multiplying the difficulty rating by the degree of success.

SECONDARY OUTCOMES:
Psychological Well-Being Scale | 18 months (3 measurements at 6-month intervals)
  An 18-item survey that measures eudaemonic well-being.
Empowerment at Work Scale | 18 months (3 measurements at 6-month intervals)
  A 12-item survey that measures a physician's sense of meaning, competence, self-determination, and impact while at work.
Abbreviated Two-Item Maslach Burnout Inventory | 18 months (3 measurements at 6-month intervals)
  A two-item survey that measures participant burnout.
Depression, Anxiety, and Stress Scale (DASS 21) | 18 months (3 measurements at 6-month intervals)
  A 21-item self-report questionnaire designed to measure the severity of the core symptoms of depression, anxiety, and stress in both clinical and nonclinical scenarios.
Leadership Self-Efficacy Scale | 18 months (3 measurements at 6-month intervals)
  A 5-item scale of leadership self-efficacy.
Self-Insight Scale | 18 months (3 measurements at 6-month intervals)
  An 8-item sub-scale of the Self-reflection and Insight Scale. This scale measures individuals' levels of insight into their thoughts, feelings and behaviors.
Solution-Focused Thinking Scale | 18 months (3 measurements at 6-month intervals)
  A 12-item scale with three subscales: Problem Disengagement, Goal Orientation, and Resource Activation.
Tolerance for Ambiguity Scale | 18 months (3 measurements at 6-month intervals)
  An eight-item assessment that measures tolerance for ambiguity.
Perspective Taking Scale | 18 months (3 measurements at 6-month intervals)
  A 7-item subscale of The Empathy Questionnaire that measures perspective-taking.
Qualitative Summary of Coaching Program | After 6-month coaching intervention. 18 months
  An open-ended interview covering issues such as 1) participant's experience with the coaching process and coach; 2) participant goals; 3) impact on the participant's workplace; 4) impact on participant's personal life; and 5) what the participant plans to do to sustain any changes or learnings.
Subject-Object Interview | 18 months
  A one-time 60 to 75-minute private interview that measures the particpant's order of subject-object development based upon constructive-developmental theory.

CONTACTS AND LOCATIONS:
Overall Officials: Richard C Winters, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided
We may make anonymized individual participant data (IPD) available to other researchers. It may be available after the completion of the trial to those who contact the PI directly.

REFERENCES:
- [Background] Theeboom, T., B. Beersma, and A.E.M. van Vianen, Does coaching work? A meta-analysis on the effects of coaching on individual level outcomes in an organizational context. The Journal of Positive Psychology, 2013. 9(1): p. 1-18.
- [Derived] Silva JAM, Mininel VA, Fernandes Agreli H, Peduzzi M, Harrison R, Xyrichis A. Collective leadership to improve professional practice, healthcare outcomes and staff well-being. Cochrane Database Syst Rev. 2022 Oct 10;10(10):CD013850. doi: 10.1002/14651858.CD013850.pub2. PMID 36214207
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials